CLINICAL TRIAL: NCT04748497
Title: Evaluation of Performance in Paralympic Athletes: Performance Outcomes in Sports
Brief Title: Performance Assessement for Paralympic Athletes
Acronym: PARAPERF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP201139; 2020-A02919-30 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-12-11; First posted 2021-02-10 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Paralympic Athletes; Sportive Performance
Keywords: paralympic athletes; performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parasportives of various disciplines (Other)
  Interventions: Other: Standardization of evaluation and follow-up

INTERVENTIONS:
Other: Standardization of evaluation and follow-up — Standardization of evaluation and clinical and sportive follow-up of athletes.
  Made-to-measure technical supports will be tested regarding the Paralympic regulations.

SUMMARY:
The primary objective of the study: improvement of sportive performances by quantification and performances monitoring of paralympic athletes.

The secondary objectives of the study:

* quantification and performances monitoring of mechanical performances during the filed tests, the laboratory analysis and the sportive competitions;
* quantification and performances monitoring of physiological performances during the filed tests, the laboratory analysis and the sportive competitions;
* quantification and risk monitoring of discipline-relative musculo-squeletic troubles, caused by training or using of sportive equipment;
* quantification and mechanical monitoring by the made-to-measure or usual sportive material.

DETAILED DESCRIPTION:
The sportive performance results from a range of determinations such as: physiological, biomechanical, morphological, psychological, social and environmental factors. The interactions between athletes, equipment, training and environment influences the development of athletes' performance. In the context of the coming Paris 2024 Paralympic Games, the performance construction for the exploration, the quantification and the management of all factors is an commun objective between sportive team, medical team and researchers.

ELIGIBILITY:
Inclusion Criteria:

* High-lever paralympic athletes registered on the ministerial list or selected by Parasport Federation of France or Shooting Federation of France;
* Aged >= 14 years;
* Informed consent signed by adult athlete or by holder of parental authority or guardian for minor athlete;
* Covered by social security system.

Exclusion Criteria:

* Temporary or definitive contraindication to the practice of the affected sport activity;
* Undergoing anti-coagulated treatments;
* Cognitive disabilities conducting impossibility to participating to clinical trial, such as serious cognitive troubles, behaviors troubles, psychic troubles or upgraded curatorship needing;
* Under guardianship or judicial decision;
* Ongoing pregnancy.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Dynamic sportive activity | through study completion, an average of 1 year
  Dynamic sportive activity: Sprint Capacity Test will be used to have maximal speed.
Dynamic sportive activity | at 42 months
  Dynamic sportive activity: Sprint Capacity Test will be used to have maximal speed.
Static sportive activity | through study completion, an average of 1 year
  Static sportive activity: maximal speed of movement of pression center.
Static sportive activity | at 42 months
  Static sportive activity: maximal speed of movement of pression center.

SECONDARY OUTCOMES:
Biomechanical indices of performance: isometric power measurement | through study completion, an average of 1 year
  Isometric power will be measured by MicroFet & handgrip of 26 measures, advice for healthcare professionals to measure handgrip strength forces to test and document grip deficits and to evaluate consistency of effort.
Biomechanical indices of performance: arms and shoulder's Strength | through study completion, an average of 1 year
  Arms and shoulder's Strength will be measured by force platform.
Physiological indices of performance: maximal aerobic speed (MAS) | Twice through study completion, an average of 42 months
  Maximal aerobic speed (MAS) will be measured by Repetition Per Minute on a Arm ergometer.
Physiological indices of performance: maximal aerobic power | Twice through study completion, an average of 42 months
  Maximal aerobic power will be measured by following Watts fluctuation during the incremental hand-biking test.
Fatigue assessment | Twice through study completion, an average of 42 months
  Fatigue assessment will be measured by Fatigue Index (Power max ratio).
Blood lactate concentration | immediately after the intervention
  Blood lactatemia level will be measured by lactometer.
VO2 peak oxygen uptake | through study completion, an average of 1 year
  VO2 peak oxygen uptake
Peak breath expiration volume assessment | through study completion, an average of 1 year
  VE peak: peak breath expiration volume
Peak cardiac frequence | through study completion, an average of 1 year
  CF: peak cardiac frequence
Musculo-squeletic troubles risks measurement | through study completion, an average of 1 year
  Musculo-squeletic troubles risks will be measured by medical following and clinical method of functional assessment of the shoulder (i.e. "Constant scale").
Time and distance of deceleration of wheelchair during riding test | through study completion, an average of 1 year
  Time and distance of deceleration of wheelchair during riding test: measured by signal analysis of instrumented wheelchair (inertial control units).
Mechanical indices of wheelchair propulsion - applied forces on handrim during the propulsion | through study completion, an average of 1 year
  Applied forces on handrim during the propulsion: measured by force platform.
Acceleration profil during the propulsion | through study completion, an average of 1 year
Speed profil during the propulsion | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: François Genêt, MD, PhD, Principal Investigator — Service Médecine Physique et de Réadaptation, Hôpital Raymond Poincaré, APHP; Jean François Toussaint, MD, PhD, Study Director — Centre d'Investigation en Médecine du Sport, Hôpital Hôtel Dieu, APHP
Locations (1):
- Service Médecine Physique et de Réadaptation, Hôpital Raymond Poincaré, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No